CLINICAL TRIAL: NCT03868995
Title: The Efficacy of Hypertonic Dextrose Injection to Anterior Talofibular Ligament Sprain: A Randomized Controlled Trial
Brief Title: The Efficacy of Hypertonic Dextrose Injection to Anterior Talofibular Ligament Sprain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N201810066
Record Dates: First submitted 2019-01-21; First posted 2019-03-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham injection (Sham Comparator): Dextrose water injection to subcutaneous layer at tender point
  Interventions: Procedure: Sham injection
- Tendon injection (Experimental): Dextrose water injection to injured tendon
  Interventions: Procedure: Tendon injection

INTERVENTIONS:
Procedure: Sham injection — Dextrose water injection to subcutaneous layer at tender point
  Arms: Sham injection
Procedure: Tendon injection — Dextrose water injection to injured tendon
  Arms: Tendon injection

SUMMARY:
Anterior talofibular ligament is the most injured ligament in ankle sprain. Investigators will include ankle sprain patients who have ankle pain or instability more than 3 months. Ultrasonography will be done for confirm ligament injury. Participants will be randomized into two groups. Participants in dextrose injection group will accept dextrose 15% injection to tendon and enthesis. In the other hand, subcutaneous sham injection to control group. Pain condition, stability test and function test, will be evaluated in 1 week, 4 weeks and 12 weeks after injection.

DETAILED DESCRIPTION:
Background: Sprains constitute most of ankle injury and 85% ankle sprain is inversion injury. The conventional treatment includes medication, physical therapy, bracing and steroid injection. Anterior talofibular ligament is the most injured ligament in ankle sprain. Although the response of acute ligament sprain is usually quickly, treatment of chronic ligament sprain is difficult. Chronic pain and ankle instability is the most common symptom in chronic ankle sprain. Dextrose prolotherapies been used for treating soft tissue injury such as osteoarthritis, tendinopathy and ligament sprain. However, there is not randomized control trial for hypertonic dextrose injection to chronic ankle sprain.

Methods: Investigators will include 40 ankle sprain patients who have ankle pain or instability sensation more than 3 months. Ultrasonography will be done for confirm ligament injury. Participants will be randomized into two groups. Dextrose injection group will accept dextrose 15% injection to tendon and enthesis. Otherwise, investigators will do subcutaneous sham injection to control group. Investigators will measure pain threshold and peak pressure by algometer, the degree of ankle instability by ultrasound, the proprioception by single leg standing, and foot and ankle questionnaire. The examination will be done before injection, immediately after injection, 1 week, 4 weeks and 12 weeks after injection.To our hypothesis, investigators suggest dextrose prolotherapy injection could decrease pain and improved proprioception.

ELIGIBILITY:
Inclusion Criteria:

1. 20-70 age
2. Chronic ankle sprain more than 3months with chronic ankle pain or instability sensation
3. Ultrasound diagnosed anterior talofibular ligament sprain

Exclusion Criteria:

1. Acute ankle sprain less than 3 months
2. Lower limb fracture history
3. Cognitive impairment
4. Other neurological or muscular disorders
5. Sever pain could not tolerate examination

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Ankle pain | Change from baseline VAS at 1 week
  visual analogue scale(VAS), range 0-10, the higher scale the worsen pain
Ankle pain | Change from baseline VAS at 4 week
  visual analogue scale(VAS), range 0-10, the higher scale the worsen pain
Ankle pain | Change from baseline VAS at 12 week
  visual analogue scale(VAS), range 0-10, the higher scale the worsen pain

SECONDARY OUTCOMES:
Ankle proprioception | Change from baseline of difference of ankle degree at 1 week
  The accuracy of ankle range of motion at 0 degree, half of dorsiflexion and half of plantar flexion
Ankle proprioception | Change from baseline of difference of ankle degree at 4 weeks
  The accuracy of ankle range of motion at 0 degree, half of dorsiflexion and half of plantar flexion
Ankle proprioception | Change from baseline of difference of ankle degree at 12 weeks
  The accuracy of ankle range of motion at 0 degree, half of dorsiflexion and half of plantar flexion
Ankle function | Change from baseline FADI at 1 week
  Foot & Ankle Disability Index (FADI), range 0-136, the higher the worse
Ankle function | Change from baseline FADI at 4 weeks
  Foot & Ankle Disability Index (FADI), range 0-136, the higher the worse
Ankle function | Change from baseline FADI at 12 weeks
  Foot & Ankle Disability Index (FADI), range 0-136, the higher the worse

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsuan Cheng, MS, Study Director — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei medical university, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided